CLINICAL TRIAL: NCT03603457
Title: OFSEP High Definition Cohort
Acronym: OFSEP HD
Status: Active, not recruiting | Type: Observational
Sponsor: EDMUS Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2018-06-28; First posted 2018-07-27 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis
Keywords: Epidemiology; Prognostic factors; Stratified medicine; Quality of life; Economic assessment
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
For neurologists and patients, it appears that one major unmet need, beside of course a cure to multiple sclerosis (MS), is to better appreciate the causal factors of disease progression, and even to obtain reliable predictive tools that could apply on the individual level and at different key moments in the disease course.

The overarching objective of the OFSEP-HD cohort is to determine prognostic factors of the evolution of disability in MS in real life, looking at disease characteristics, care practices potentially modifying the evolution of the disease since MS clinical onset and along specific post-onset landmarks. This general framework leads to study 3 specific research objectives:

1. To identify determinants (socio-demographic characteristics, clinical characteristics, health related quality of life (QoL), changes in classification, and biomarkers) for the progression of MS disease and its consequences;
2. To study the effectiveness of treatments in real life;
3. To merge both determinants and treatments for creating patient-centered prognostic tools for identifying specific subgroups of patients and helping making decision to start, maintain or adapt care management.

To achieve these objectives, the OFSEP (The French multiple sclerosis registry) infrastructure, managed under a quality insurance system, offers a unique opportunity for the first time in France to create a large cohort of MS cases, providing high-definition and sequential multimodal data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis according to the most recent criteria at entry into the HD cohort
* Followed in one MS Clinical Reference Centre (CRC SEP)
* Newly diagnosed after the study start or
* If MS onset occurred before study start, regular follow-up in a CRC SEP
* Irreversible disability ≤ 7.0 (permanent use of a wheelchair) on EDSS at inclusion in the study

Non-inclusion Criteria:

* Inability to answer questionnaires
* Pregnant women at the time of inclusion

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All MS patients from MS Clinical Reference Centre (CRC SEP).
Sampling Method: Non-Probability Sample
Enrollment: 2842 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to reach irreversible Expanded Disability Status Scale (EDSS) scores of 6 | Through study completion, an average of 2 years
Activity of disease | 1 year
  Activity is determined, according Lublin 2014, by clinical relapses and/or MRI activity (contrast-enhancing lesions ; new or unequivocally enlarging T2 lesions assessed at least annually)
Change in T2 lesion load evaluated by analysis of raw MRI | 1 year
Change in quality of life evaluated by EQ-5D-5L scale | 1 year
  The 5-level EQ-5D version (EQ-5D-5L) consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The five dimensions can be combined into a number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Change in quality of life evaluated by SF-12 scale | 1 year
  The SF-12 questionnaire uses 12 questions to measure functional health and well-being from the patient's point of view.
Change in quality of life evaluated by MusiQoL scale | 1 year
  The MusiQoL (Multiple Sclerosis International Quality of Life Questionnaire) is a multidimensional Health Related Quality of Life instrument that provides information based on the views and perceptions of the participants.

CONTACTS AND LOCATIONS:
Locations (25):
- France (24):
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Créteil, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - CHU Pitié-Salpétrière, Paris
  - CHU Saint-Antoine, Paris
  - Fondation Rothschild, Paris
  - CHI de Poissy-Saint-Germain-en-Laye, Poissy
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours
- CHU de Fort-de-France, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Yes
URL: http://www.ofsep.org/en/data-access

REFERENCES:
- [Derived] Guillemin F, Casey R, Epstein J, Foucher Y, Laplaud D, Achit H, Rollot F, Leray E, Vukusic S; OFSEP-HD investigators. Prognostic factors of disability progression in multiple sclerosis in real life: the OFSEP-high definition (OFSEP-HD) prospective cohort in France. BMJ Open. 2025 Apr 7;15(4):e094688. doi: 10.1136/bmjopen-2024-094688. PMID 40194873